CLINICAL TRIAL: NCT06544993
Title: Evaluation of the Efficacy and Safety of Microneedling Combined With Botulinum Toxin-A Versus Meso-Botox Injection in the Treatment of Atrophic Acne Scars: A Split-face Comparative Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mariam Nashaat latif, Resident AT DERMATOLOGY department-sohag general hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soh-Med-24-07-21MS
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Atrophic Acne Scar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- right side of face (Active Comparator): meso-Botox injection
  Interventions: Drug: Meso-botox
- left side of face (Active Comparator): microneedling combined with Botulinum toxin-A
  Interventions: Drug: Meso-botox

INTERVENTIONS:
Drug: Meso-botox — Micro-Botox, is a highly diluted Botulinum toxin type A
  Other Names: Micro-Botox

SUMMARY:
Post-acne scars are psychologically disappointing and therapeutically challenging condition. No standard treatment for atrophic acne scars.

Micro-Botox, is a highly diluted BTX-A which could be injected safely intra-dermally. It targets the superficial fibers of facial muscles, sweat, and sebaceous glands inducing pores shrinkage, decreasing the sebum and excessive sweating, in addition to face lifting and reducing fine wrinkles without affecting emotions, this subsequently makes the skin tighter and gives the facial skin a smooth appearance.

Also, BTX-A appears to have an inhibitory effect on fibroblasts and collagen remodeling activity, in addition to releasing muscular tension at scar edges through superficial muscle relaxation. So, it can reduce the tethering and pulling effect of the muscles surrounding the acne scars. Also, it has anti-inflammatory and angiogenesis induction effects. Therefore, micro-Botox is believed to improve acne scars.

Therefore, it will be interesting to compare the efficacy and safety of microneedling combined with BTX-A versus meso-Botox injection in the treatment of atrophic acne scars through a split-face clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrophic post-acne scars.

Exclusion Criteria:

* Pregnancy and lactation. Ongoing infection within the targeted treatment region or active acne lesions. Skin cancer, or precancerous lesions. History of keloid formation. History of allergy to BTX. Patients with neuromuscular diseases, patients with pre-existing medical conditions that cause muscle weakness as myasthenia gravis.

Patients who underwent Botox injection, during the last 6 months. Patients who were under treatment by systemic retinoids in the previous 6 months.

Patients with a history of chemical peels or laser procedures within 6 months of the study period.

Patients with bleeding disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Goodman and Baron Qualitative Global Scarring Grading System: | 6 months
  Acne scarring severity will be graded before and after treatment. Grade 1 (macular) erythematous, hyper/hypopigmented flat marks; Grade 2 (mild) mild atrophy or hypertrophic scars that may not be obvious at a distance of 50cm or greater & may be covered adequately by makeup or beard hair in men; Grade 3 (moderate) moderate atrophy or hypertrophic scarring obvious at a distance of 50cm or greater, not covered by makeup or beard hair but can be flattened by manual stretching of the skin; and Grade 4 (severe) severe atrophy or hypertrophic scarring not flattened by manual stretching of the skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mohamed NE, Shabaan SN, Raouf AH. Microbotox (Mesobotox) versus microneedling as a new therapeutic modality in the treatment of atrophic post-acne scars. J Cosmet Dermatol. 2022 Dec;21(12):6734-6741. doi: 10.1111/jocd.15419. Epub 2022 Oct 14. PMID 36169570
- [Background] Fabi SG, Park JY, Goldie K, Wu W. Microtoxin for Improving Pore Size, Skin Laxity, Sebum Control, and Scars: A Roundtable on Integrating Intradermal Botulinum Toxin Type A Microdoses Into Clinical Practice. Aesthet Surg J. 2023 Aug 17;43(9):1015-1024. doi: 10.1093/asj/sjad044. PMID 36857534
- [Background] Jung JH, Jin SG. Microneedle for transdermal drug delivery: current trends and fabrication. J Pharm Investig. 2021;51(5):503-517. doi: 10.1007/s40005-021-00512-4. Epub 2021 Mar 4. PMID 33686358
- [Background] Ebrahim H, Elardi A, Khater S, Morsi H. Successful Topical Application of Botulinum Toxin After Microneedling Versus Microneedling Alone for the Treatment of Atrophic Post Acne Scars: A Prospective, Split-face, Controlled Study. J Clin Aesthet Dermatol. 2022 Jul;15(7):26-31. PMID 35942010